CLINICAL TRIAL: NCT04395833
Title: Emerging Health Challenges for Children With Motor Disabilities and Their Parents Facing the COVID-19 Pandemic: Messages From Families Answering the ECHO French National Survey
Brief Title: National Survey on the Lockdown of Children With Disabilities
Acronym: ECHO
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: CHRU de BREST ECHO
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Identify Emerging Health Challenges for Children With Motor Disabilities and Their Parents Facing the COVID-19 Pandemic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During the COVID-19 pandemic, lockdown measures were established in France affecting the life course of children with disabilities. This study aimed at identifying the experiences, main difficulties and needs of these children and their parents during the lockdown period.

ELIGIBILITY:
Inclusion Criteria:

-children (age 0-18 years) with motor disabilities (with and without associated impairement), living in France.

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with motor disabilities, with and without associated impairement
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Experience during lockdown | From the 6th of April 2020 until the 11th of May 2020
  Identify the lived experience, the needs, and difficulties of children with motor disabilities and their parents during the COVID-2019 lockdown
Health risk during lockdown | From the 6th of April 2020 until the 11th of May 2020
  Identify the risks on health of children with motor disabilities due to the COVID-2019 lockdown
Impact on medical and rehabilitation follow up | From the 6th of April 2020 until the 11th of May 2020
  Identify the impact on the medical and rehabilitation follow up of children with disabilities during COVID-19 lockdown
Impact on daily living | From the 6th of April 2020 until the 11th of May 2020
  Identify the impact on the daily living of children with motor disabilities and their families during the COVID-19 lockdown

SECONDARY OUTCOMES:
Experience during lockdown | From the 24th of April 2020 until the 11th of May 2020
  Identify the lived experience, the needs, and difficulties of children without motor disabilities and their parents during the COVID-2019 lockdown

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France